CLINICAL TRIAL: NCT04150276
Title: Zero Positive End-expiratory Pressure Before Emergence Improves Postoperative Oxygenation in Obese Patients Undergoing Laparoscopic Surgery - a Randomized Clinical Trial
Brief Title: Obesity, PEEP and Postoperative Oxygenation
Acronym: ZAPPAII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Västmanland (Other)
Responsible Party: Principal Investigator, Erland Ostberg, Consultant, principal investigator, Region Västmanland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Dnr 2019/04860
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Oxygenation
Keywords: Oxygenation; Positive end-expiratory pressure; General anaesthesia; Obesity; Atelectasis; Mechanical ventilation
MeSH Terms: conditions — Obesity; Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZEEP during awakening (Active Comparator): ZEEP will be used during emergence preoxygenation and awakening.
  Interventions: Procedure: ZEEP during awakening
- PEEP during awakening (Active Comparator): PEEP is maintained throughout emergence preoxygenation and awakening.
  Interventions: Procedure: PEEP during awakening

INTERVENTIONS:
Procedure: ZEEP during awakening — ZEEP will be established 2 min prior to the start of emergence preoxygenation and awakening.
  Arms: ZEEP during awakening
Procedure: PEEP during awakening — PEEP will be maintained throughout emergence preoxygenation and awakening.
  Arms: PEEP during awakening

SUMMARY:
A study on overweight patients undergoing anesthesia for laparoscopic surgery.

- evaluation of positive end-expiratory pressure versus zero positive end-expiratory pressure during awakening on oxygenation in the early postoperative period.

DETAILED DESCRIPTION:
Positive end-expiratory pressure (PEEP) is often used during mechanical ventilation to preserve end-expiratory lung volume. After emergence and extubation, this volume will diminish instantly. Some patients will have difficulties to restore functional residual capacity (FRC) during the early phase of recovery. If routine high FIO2 is being delivered together with maintained PEEP prior to extubation, several important prerequisites are established for the development of postoperative atelectasis. The investigators hypothesize that establishing zero positive end-expiratory pressure (ZEEP) immediately prior to emergence preoxygenation, will prevent gas with high oxygen concentration from entering dorso-basal areas of the lungs, and thereby diminishing postoperative atelectasis formation and improve oxygenation.

This randomized controlled study will study overweight patients undergoing general anesthesia for laparoscopic surgery. The patients in the two study groups will receive mechanical ventilation with identical settings, comprising low TV, PEEP, and no RM. Randomization will occur at the end of surgery, before awakening. The patients will be allocated to zero PEEP (ZEEP) or maintained PEEP during emergence preoxygenation and extubation. Importantly, the intervention group will have ZEEP established while still having low ETO2 levels, prior to any preoxygenation. Arterial blood gases will be collected before, during and after anaesthesia. Primary endpoint measure will be change in oxygenation from before awakening to after awakening.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients scheduled for elective laparocopic surgery.
* American Society of Anesthesiologists functional class I-III
* Body Mass Index 35-50 kg/m2

Exclusion Criteria:

* Body Mass Index ≥50 kg/m2
* Peripheral oxygen saturation (SpO2) breathing air <94 %
* Symtomatic asthma, COPD or heart failure
* Ischemic heart disease
* Hemoglobin < 100g/l
* Smokers and ex-smokers that stopped smoking < 9 months ago
* Need for peroperative RM and PEEP higher than in study protocol, as indicated by SpO2 <92% despite the stipulated FiO2 0.30-0.35.
* Obstructive sleep apnea syndrome on home-CPAP

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Change in oxygenation | Bloodgases will be obtained 5 minutes before the start of the awakening procedure and 30 minutes after awakening and extubation.
  Arterial blood samples will be collected for measurement of arterial oxygen partial pressure.

SECONDARY OUTCOMES:
Need for postoperative supplemental oxygen | First 3 hours postoperatively.
  Number of patients and amount of oxygen needed in the respective group postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Erland Östberg, MD, PhD, Principal Investigator — Region Västmanland
Locations (1):
- Dep. of Anaesthesia and Intensive Care, Västerås, Region Västmanland, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Please email request to the study principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after publication of study results, approximately 18 months after study completion.
Access Criteria: Data access requests will be reviewed by a review panel at the Center for Clinical Research, Västerås. Requestors will be required to sign a data acess agreement.

REFERENCES:
- [Derived] Ostberg E, Larsson A, Wagner P, Eriksson S, Edmark L. Positive end-expiratory pressure and emergence preoxygenation after bariatric surgery: effect on postoperative oxygenation: A randomised controlled trial. Eur J Anaesthesiol. 2025 Jan 1;42(1):54-63. doi: 10.1097/EJA.0000000000002071. Epub 2024 Oct 3. PMID 39325031